CLINICAL TRIAL: NCT06917989
Title: Evaluation of the Effect of Relaxation Exercise and Virtual Reality Application on Pain, Trismus, Sleep, Kinesiophobia and Anxiety Level After Impacted Third Molar Dental Surgery
Brief Title: Evaluation of the Effect of Relaxation Exercise and Virtual Reality Application After Impacted Third Molar Dental Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Emre Serdar Atalay, Assistant Professor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/001; Academician (Other: University of Health Sciences Türkiye)
Record Dates: First submitted 2025-03-28; First posted 2025-04-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Virtual Reality; Relaxation; Third Molar Surgery; Pain
Keywords: Virtual Reality; Relaxation; Third Molar Surgery; Pain
MeSH Terms: conditions — Pain | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Group 1 will be given a Relaxation Exercise, Group 2 will be given a Virtual Reality Application in Addition to the Relaxation Exercise. Group 3 will be the control group. Patient education will be given to all groups as Group 1, Group 2 and Group 3. Participants will be between the ages of 18-35.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Relaxation Exercise (Experimental): Consist of participants who underwent Relaxation Exercise and Patient Education
  Interventions: Other: Relaxation Exercise; Other: Patient Education
- Virtual Reality Application in Addition to the Relaxation Exercise (Experimental): Consist of participants who underwent Relaxation Exercise and Virtual Reality Application and Patient Education
  Interventions: Other: Relaxation Exercise; Other: Virtual Reality Application; Other: Patient Education
- Control Group (Other): Consist of participants who underwent Patient Education
  Interventions: Other: Patient Education

INTERVENTIONS:
Other: Relaxation Exercise — Jacobson muscle relaxation technique
  Arms: Relaxation Exercise; Virtual Reality Application in Addition to the Relaxation Exercise
Other: Virtual Reality Application — Virtual Reality Application will be done using virtual reality glasses
  Arms: Virtual Reality Application in Addition to the Relaxation Exercise
Other: Patient Education — Participants will be informed about oral care, food consumption, nutrition and sleeping position.

SUMMARY:
Impacted tooth extractions are the most frequently performed procedure in oral surgery. Complications such as pain and trismus are frequently observed after surgery. Pain, especially after surgery, causes serious discomfort to the individual. These complications negatively affect the daily lives of individuals. Decreased sleep quality, increased anxiety, fear of moving the jaw joint, decreased quality of life, and loss of labor are among the examples that can be given. It is important for individuals to have a more comfortable process in the early period after surgery. During this period, individuals receive pharmacological treatment; however, non-pharmacological approaches should not be ignored. Evaluation of the effects of relaxation exercise and virtual reality application applied after impacted third molar surgery on pain, trismus, sleep, kinesiophobia, and anxiety levels.

DETAILED DESCRIPTION:
Impacted third molar surgery is one of the most common procedures performed by oral, dental and maxillofacial surgeons. During surgical removal of teeth, trauma may occur due to the narrowing of the area and insufficient visibility, the position of the teeth and the hardness of the bone structure. In addition, this surgical procedure leads to various complications since it requires intraoral intervention. It has also been stated that most complications are triggered by the inflammatory process after surgery and are reported with varying frequencies. As a result of trauma that may occur in soft and bone tissue, symptoms such as pain, swelling and trismus may occur. Post-surgical pain is an acute type of pain that begins with surgical trauma, gradually decreases and ends with tissue healing. This pain triggers a stress response in the sympathetic nervous system, causing an increase in muscle tension. Another situation encountered after surgery is an increase in anxiety. Anxiety is a distinct state of restlessness caused by fear, distress or apprehension. Individuals are afraid of surgery even if they think surgery is necessary to regain their health or improve their quality of life. The incidence of complications is higher in individuals with high levels of anxiety after surgery.

In the evaluation; Modified Dental Anxiety Scale, Visual Analog Scale, Maximum Active Mouth Opening Measurement, The Tampa Scale for Kinesiophobia for Temporomandibular Disorders, Electromyography (EMG), Turkish version of the Visual Analog Sleep Scale, State and Trait Anxiety Scale will be used.

Individuals participating in the study will be included in one of 3 groups. Group 1 will be Relaxation Exercise, Group 2 will be Virtual Reality Application in addition to Relaxation Exercise, and Group 3 will be the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* According to the Pell and Gregory classification; Having undergone surgery on a mandibular third molar with Class 2-3, Position B and C impaction degree
* Being systemically healthy (ASA 1)
* Not having high dental anxiety according to the Modified Dental Anxiety Scale (<19)
* Individuals who have undergone bone removal during surgery
* Individuals who do not have any psychiatric problems
* Presence of pain <3 months

Exclusion Criteria:

* Presence of myofascial pain affecting the temporomandibular joint
* Presence of tumoral structure related to the impacted third molar
* Presence of acute pericoronitis
* Presence of bruxism
* Presence of vertigo, seizures, epilepsy, active nausea and vomiting
* Having a beard but not preferring to shave (shaved skin is required for accurate EMG measurement)
* Pregnancy
* Smoking and alcohol addiction
* Individuals with sleep disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Dental Anxiety | Before impacted third molar extraction
  Modified Dental Anxiety Scale: The lowest total score to be received on the entire survey is 5, the highest score is 25. A high score denoted a high anxiety response.
Pain Level | Before the impacted third molar extraction - within 30 minutes after impacted third molar extraction - post-operative 2nd and 7th day
  Visual Analog Scale: At the left end of the scale (0 cm) is "no pain"; at the right end (10 cm) is "worst pain". (0: no pain, 10: unbearable pain). The higher the score, the higher the pain level.
Maximum Active Mouth Opening | Before the impacted third molar extraction - within 30 minutes after impacted third molar extraction - post-operative 2nd and 7th day
  Therabite Range of Motion Scale: According to the measurement results made with the ruler, the value obtained will increase as the mouth opening distance increases.
Kinesiophobia Level | Before the impacted third molar extraction - within 30 minutes after impacted third molar extraction - post-operative 2nd and 7th day
  The Tampa Scale for Kinesiophobia for Temporomandibular Disorders: 12-48 points are received on this scale. The higher the score the person receives, the higher the level of kinesiophobia
Muscle Activity | Before the impacted third molar extraction - within 30 minutes after impacted third molar extraction - post-operative 2nd and 7th day
  Electromyography
Sleep Quality | Before the impacted third molar extraction - within 30 minutes after impacted third molar extraction - post-operative 2nd and 7th day
  Turkish version of the Visual Analog Sleep Scale: The scale is scored between 0 and 1000. The higher the score received from the scale indicates that the quality of sleep has decreased.
Anxiety Level | Before the impacted third molar extraction - within 30 minutes after impacted third molar extraction - post-operative 2nd and 7th day
  State-Trait Anxiety Inventory: The highest score is 80, the lowest score is 20. The higher the total anxiety score, the higher the anxiety level of the person filling out the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ju W, Ren L, Chen J, Du Y. Efficacy of relaxation therapy as an effective nursing intervention for post-operative pain relief in patients undergoing abdominal surgery: A systematic review and meta-analysis. Exp Ther Med. 2019 Oct;18(4):2909-2916. doi: 10.3892/etm.2019.7915. Epub 2019 Aug 19. PMID 31555379
- [Background] Georgescu RD, Dobrean A, Silaghi CA, Silaghi H. A virtual reality-based intervention for surgical patients: study protocol of a randomized controlled trial. Trials. 2021 Apr 19;22(1):289. doi: 10.1186/s13063-021-05196-7. PMID 33874974
- [Background] Gurram P, Narayanan V, Chandran S, Ramakrishnan K, Subramanian A, Kalakumari AP. Effect of Heartfulness Meditation on Anxiety and Perceived Pain in Patients Undergoing Impacted Third Molar Surgery. J Oral Maxillofac Surg. 2021 Oct;79(10):2060.e1-2060.e7. doi: 10.1016/j.joms.2021.04.027. Epub 2021 Apr 29. PMID 34097862
- [Background] Topcu SY, Findik UY. Effect of relaxation exercises on controlling postoperative pain. Pain Manag Nurs. 2012 Mar;13(1):11-7. doi: 10.1016/j.pmn.2010.07.006. Epub 2010 Sep 21. PMID 22341136